CLINICAL TRIAL: NCT07012551
Title: Endovascular Modalites for Contralateral Common Iliac Artery in Patients With Symptomatic Unilateral Common Iliac Artery Occlusive Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Shawki Roshdi, assistant lecturer, Assiut University
Other Study IDs: Common iliac artery stenting
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Iliac Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Common iliac artery stenting — Stenting of common iliac artery by balloon mounted stent

SUMMARY:
To evaluate the safety, efficacy, and outcomes of endovascular strategies for protection of the contralateral CIA in patients with symptomatic unilateral CIA occlusive disease

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients (Rutherford category 3- 5) due to Unilateral common iliac artery occlusive disease.

with or without combined iliac or femoropopliteal or infrapopliteal lesions.

Asymptomatic Contralateral limb.

Patent at least one run-off vessel

Exclusion Criteria:

* Distal aorta lesion

contralateral CIA occlusion

Previous endovascular or surgical procedures for the same lesion

Hypersensitivity to contrast material

Presence of aortic or iliac aneurysms

Patients with unsalvageable limb

Non atherosclerotic lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the Vascular Surgery Clinics in Assiut University Hospitals complaining of unilateral CIA ostial occlusive disease, Rutherford category 3, 4and 5 will be recruited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency of both common iliac arteries | 2 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboyans V, Desormais I, Lacroix P, Salazar J, Criqui MH, Laskar M. The general prognosis of patients with peripheral arterial disease differs according to the disease localization. J Am Coll Cardiol. 2010 Mar 2;55(9):898-903. doi: 10.1016/j.jacc.2009.09.055. PMID 20185041